CLINICAL TRIAL: NCT00317915
Title: The Irbesartan in Patients With Type 2 Diabetes and Microalbuminuria (IRMA 2)
Brief Title: Irbesartan in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Bristol-Myers Squibb (Industry); Sanofi-Synthelabo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC2481
Record Dates: First submitted 2006-04-24; First posted 2006-04-25 (Estimated); Last update posted 2006-04-25 (Estimated); Status verified 2006-04

CONDITIONS: Type 2 Diabetes; Microalbuminuria; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

INTERVENTIONS:
Drug: Irbesartan treatment

SUMMARY:
The aim of this multicenter, doubleblind, randomized study was to investigate the renoprotective effect of irbesartan treatment in patients with type 2 diabetes and microalbuminuria (a precursor of diabetic kidney disease). 590 patients were randomized to a median 24 months of treatment with 300 mg irbesartan once daily, 150 mg irbesartan once daily or placebo. Time to development of overt nephropathy, defined by persistent proteinuria, was the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes. Hypertension. Persistent microalbuminuria. Serum creatinine concentration of no more than 1.5 mg per deciliter (133 µmol per liter) for men and no more than 1.1 mg per deciliter (97 µmol per liter) for women. -

Exclusion Criteria:

Nondiabetic kidney disease. Cancer. Life-threatening disease with death expected to occur within two years. Indication for angiotensin-converting- enzyme (ACE) inhibitors or angiotensin-II-receptor antagonists. -

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Development of overt nephropathy

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Henrik Parving, Prof. DMsc, Principal Investigator — Steno Diabetes Center Copenhagen

REFERENCES:
- [Derived] Jongs N, Gasparyan SB, Frison L, Schloemer P, Brinker M, Little DJ, Heerspink HJL. Use of eGFR Slope Thresholds as End Point Components in a Kidney Disease Progression Hierarchical Composite End Point. J Am Soc Nephrol. 2025 Dec 1;36(12):2421-2430. doi: 10.1681/ASN.0000000766. Epub 2025 Jun 17. PMID 40526444
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Heerspink HJL, Jongs N, Schloemer P, Little DJ, Brinker M, Tasto C, Karpefors M, Wheeler DC, Bakris G, Perkovic V, Nkulikiyinka R, Rossert J, Gasparyan SB. Development and Validation of a New Hierarchical Composite End Point for Clinical Trials of Kidney Disease Progression. J Am Soc Nephrol. 2023 Dec 1;34(12):2025-2038. doi: 10.1681/ASN.0000000000000243. Epub 2023 Oct 24. PMID 37872654
- [Derived] Piazza M, Hanssen NMJ, Persson F, Scheijen JL, van de Waarenburg MPH, van Greevenbroek MMJ, Rossing P, Hovind P, Stehouwer CDA, Parving HH, Schalkwijk CG. Irbesartan treatment does not influence plasma levels of the dicarbonyls methylglyoxal, glyoxal and 3-deoxyglucosone in participants with type 2 diabetes and microalbuminuria: An IRMA2 sub-study. Diabet Med. 2021 Sep;38(9):e14405. doi: 10.1111/dme.14405. Epub 2020 Oct 16. PMID 32961617
- [Derived] Persson F, Rossing P, Hovind P, Stehouwer CD, Schalkwijk CG, Tarnow L, Parving HH. Endothelial dysfunction and inflammation predict development of diabetic nephropathy in the Irbesartan in Patients with Type 2 Diabetes and Microalbuminuria (IRMA 2) study. Scand J Clin Lab Invest. 2008;68(8):731-8. doi: 10.1080/00365510802187226. PMID 18609080